CLINICAL TRIAL: NCT06323018
Title: Effects of Remote Ischaemic Preconditioning in Cemented Total Hip Arthroplasty: Randomized Controlled Trial
Brief Title: Effects of Remote Ischaemic Preconditioning in Cemented Hip Arthroplasty.
Acronym: PRINCIPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Kaspar Tootsi, Principal Investigator, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 384T-26
Record Dates: First submitted 2024-03-13; First posted 2024-03-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Hip; Cardiovascular Diseases; Bone Cement Implantation Syndrome; Kidney Diseases
MeSH Terms: conditions — Osteoarthritis, Hip; Cardiovascular Diseases; Kidney Diseases | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization and intervention is done by a dedicated study nurse. Patient, orthopedic surgeon, investigator and outcomes assessor and statistician are all blinded to the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): SHAM procedure is done one hour before cemented hip arthroplasty and comprises of 4 cycles of 5min sham procedure. Everything apart from the pressure in the cuff is similar to the RIPC procedure.
  Interventions: Other: SHAM
- Remote Ischemic preconditioning group (Active Comparator): RIPC procedure is done one hour before cemented hip arthroplasty and comprises of 4 ischemia (using brachial cuff with suprasystolic blood pressure for 5 min) and reperfusion (5 min) cycles.
  Interventions: Procedure: Remote Ischemic Preconditioning

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — 4 cycles of 5 min pressure (produces an ischemia episode in subject's upper limb) with AutoRIC device (Starfish Medical, Canada)
  Arms: Remote Ischemic preconditioning group
Other: SHAM — 4 cycles of 5min light pressure (no ischemia produced) with AutoRIC device (Starfish Medical, Canada) to imitate the RIPC procedure
  Arms: Control group

SUMMARY:
Total joint arthroplasty is one of the best treatment options for end-stage osteoarthritis. Cemented hip arthroplasty is mainly indicated for elderly patients with poor bone quality and multiple comorbidities. Bone cement implantation syndrome is associated with cemented hip arthroplasty and it has been shown to increase cardiovascular and renal complication and brain damage postoperatively. The aim of this project is to elucidate whether remote-ischemic preconditioning (RIPC) has multi-organ protective effect in cemented hip arthroplasty patients.

DETAILED DESCRIPTION:
Total joint arthroplasty is one of the best treatment options for end-stage osteoarthritis. Cemented hip arthroplasty is mainly indicated for elderly patients with poor bone quality and multiple comorbidities. Cemented hip arthroplasty is strongly associated with bone cement implantation syndrome (BCIS). It is characterized by hypoxia, hypotension and/or unexpected loss of consciousness occurring around the time of cementation, prosthesis insertion or reduction of the joint. It has been shown to increase cardiovascular and renal complication and brain damage postoperatively. Remote-ischemic preconditioning has shown kidney, myocardial and brain injury protective effect on non-cardiac surgery patients. The aim of this project is to elucidate whether remote-ischemic preconditioning (RIPC) has multi-organ protective effect in cemented hip arthroplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* age >65 years
* undergoing total hip cemented hip arthroplasty

Exclusion Criteria:

* previously diagnosed peripheral artery disease on both upper limb
* RIPC is contraindicated

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury | From enrollment to 3. postoperative day
  Peak hs-cTnT value
  * baseline characteristics are measured before surgery
  * measuring is repeated 1h after surgery and up to 3 days postoperatively

SECONDARY OUTCOMES:
Cardiovascular injury | From enrollment to 3. postoperative day
  Change in baseline of hs-cTnT and NT-proBNP
  * baseline characteristics are measured before surgery
  * measurements are repeated 1h after surgery and up to 3 days postoperatively (once a day)
Clinical serious complications | From enrollment to 1 year postoperatively
  Mortality, Bone cement implantation syndrome, serious cardiovascular complications (heart attack, heart failure, stroke, arrhythmia, peripheral artery thrombosis)
  * data is collected trough Estonian National Health database "Digilugu"
  * blood pressure, saturation and patient's mental state are monitored during the operation to register any case of bone cement implantation syndrome
Carotid-femoral pulse velocity | From enrollment to 1. postoperative day
  Measured with Sphygmocor XCEL
  * baseline characteristics are measured before surgery
  * measuring is repeated 24 h after surgery
Augmentation index | From enrollment to 1. postoperative day
  Measured with Sphygmocor XCEL
  * baseline characteristics are measured before surgery
  * measuring is repeated 24 h after surgery
Brain injury | From enrollment to 3. postoperative day
  Change in baseline of S-100B and NSE
  * baseline characteristics are measured before surgery
  * measuring is repeated 1h after surgery and up to 3 days postoperatively
  Change in baseline of Choice-reaction test results done pre-and postoperatively
  * baseline test result is measured before surgery
  * measuring is repeated 24h after surgery
Kidney Injury | From enrollment to 3. postoperative day
  Change in baseline of creatinine and cystatin C
  * baseline characteristics are measured before surgery
  * measuring is repeated 1h after surgery and up to 3 days postoperatively
Total antioxidative capacity (TAC) | From enrollment to 3. postoperative day
  Change in baseline of total antioxidant capacity (TAC)
  * baseline characteristics are measured before surgery
  * measuring is repeated 1h after surgery and up to 3 days postoperatively
Oxidative stress level (total peroxide levels) | From enrollment to 3. postoperative day
  Change in baseline total peroxide levels (TPX)
  * baseline characteristics are measured before surgery
  * measuring is repeated 1h after surgery and up to 3 days postoperatively
Inflammation level | From enrollment to 3. postoperative day
  Change in baseline of inflammation markers (HIF1α, IL6, IL-1β, TNF-α, IL-10)
  * baseline characteristics are measured before surgery
  * measuring is repeated 1h after surgery and on the first postoperative day
Low molecular weight metabolites (uM) | From enrollment to 1. postoperative day
  Change in baseline of:
  Acylcarnitines Phosphatidylcholines Lysophosphatidylcholines Sphingomyelins Ceramides Dihydroceramides Hexosylceramides Dihexosylceramides Trihexosylceramides Cholesteryl esters Diglycerides Triglycerides Amino acids Amino acid related Bile acids Biogenic amines Carboxylic acids Fatty acids Hormones Indoles and derivatives

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tartu, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernits K, Martson A, Kals J, Tagoma A, Maasalu K, Aus A, Vent K, Tootsi K. Remote ischaemic preconditioning in cemented hip arthroplasty (the PRINCIPAL study)-randomised controlled trial: study protocol. BMJ Open. 2025 Jun 23;15(6):e096433. doi: 10.1136/bmjopen-2024-096433. PMID 40550717